CLINICAL TRIAL: NCT02913300
Title: Comparison of 1% Versus 2% Lignocaine for Topical Anaesthesia in Endobronchial Ultrasound Guided Transbronchial Needle Aspiration
Brief Title: 1% vs. 2 % Lignocaine for Endobronchial Ultrasound Guided Transbronchial Needle Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr. Karan Madan, MD, DM Assistant Professor, Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Lignocaine EBUS RCT
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Bronchopulmonary Diseases
Keywords: Lignocaine
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 % Lignocaine (Active Comparator): 1 % Lignocaine administered for topical anaesthesia during EBUS-TBNA
  Interventions: Drug: Lignocaine 1% concentration solution
- 2 % Lignocaine (Active Comparator): 2 % Lignocaine administered for topical anaesthesia during EBUS-TBNA
  Interventions: Drug: Lignocaine 2% concentration solution

INTERVENTIONS:
Drug: Lignocaine 1% concentration solution
  Arms: 1 % Lignocaine
Drug: Lignocaine 2% concentration solution
  Arms: 2 % Lignocaine

SUMMARY:
Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS -TBNA) is commonly performed for diagnosis of mediastinal pathologies. The procedure can either be performed under general anaesthesia or under moderate sedation with topical anaesthesia. Most patients tolerate the procedure well although cough is often reported as a distressing symptom. Topical lignocaine is administered during bronchoscopy for local anaesthesia. There is no literature on the efficacy of lower concentrations (1%) versus a higher (2%) during EBUS TBNA. This study would help to determine whether 1% lignocaine is as effective as 2% lignocaine for airway anaesthesia during EBUS-TBNA.

DETAILED DESCRIPTION:
For all patients meeting the inclusion criteria, the demographic profile including age, sex, weight, smoking history shall be recorded. A written informed consent will be obtained from all participants. The patients who undergo EBUS-TBNA under moderate sedation would be randomised in a one is to one ratio either to 1% lignocaine or 2% lignocaine group. Prior to EBUS-TBNA, Blood pressure, pulse rate, respiratory rate and pulse oximetry saturation will be recorded at the baseline Patients in both the groups shall be prepared in a similar fashion except for the concentration of lignocaine used. Two different concentration of lignocaine solution will be labelled as solution 'A' or solution 'B' containing either of 1% or 2% lignocaine solution .Operator will be provided either solution A or B based on the initial randomisation.

During the procedure, 1.5ml aliquots of the provided lignocaine solution will be delivered through the bronchoscope using spray-as-you go technique. The total number of aliquots used during the procedure will be recorded. The patients would be monitored for any adverse effects throughout the procedure. The bronchoscopist doing the procedure will be provided 2 VAS charts to mark the severity of cough and overall procedure satisfaction.

Post procedure, patients will record the pain experienced while undergoing the procedure on the faces pain rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Indication for diagnostic or therapeutic flexible bronchoscopy
* Age > 18 years

Exclusion Criteria:

* Refusal of consent
* Known documented hypersensitivity to lignocaine
* Procedure performed under general anaesthesia
* Pregnancy
* Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Operator rated cough VAS | At study completion approximately 6 months
Operator rated overall procedure satisfaction VAS | At study completion approximately 6 months

SECONDARY OUTCOMES:
Total lignocaine dose administered | At study completion approximately 6 months
Patient facies pain rating scale | At study completion approximately 6 months
Procedure related adverse events | At study completion approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, MD, DM, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided